CLINICAL TRIAL: NCT03597399
Title: A Post-Authorization, Multicenter, Longitudinal, Observational Safety Registry Study for Patients Treated With Voretigene Neparvovec in US
Brief Title: A Patient Registry Study for Patients Treated With Voretigene Neparvovec in US
Status: Completed | Type: Observational
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SPKRPE-PASS
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Confirmed Biallelic RPE65 Mutation-associated Retinal Dystrophy
Keywords: Leber Congenital Amaurosis (LCA); Inherited Retinal Dystrophy; RPE65; Retinitis Pigmentosa (RP)
MeSH Terms: conditions — Leber Congenital Amaurosis; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Biological: AAV2-hRPE65v2,voretigene neparvovec-rzyl — Subretinal administration of gene therapy vector AAV2-hRPE65v2 (voretigene neparvovec-rzyl) to both eyes via surgical procedures on separate days.
  Other Names: AAV2-hRPE65v2; voretigene neparvovec; gene therapy vector

SUMMARY:
The objective of this study is to collect long-term safety information (i.e., for 5 years after treatment) associated with voretigene neparvovec-rzyl (vector and/or transgene), its subretinal injection procedure, the concomitant use of corticosteroids, or a combination of these procedures and products.

The enrollment period will last for two years from the first treatment following product approval (through 31March2020) and include a minimum of 40 patients.

DETAILED DESCRIPTION:
Voretigene neparvovec-rzyl is a gene therapy intended for use in individuals with confirmed biallelic RPE65 mutation-associated retinal dystrophy and viable retinal cells. Mutations in the RPE65 gene are associated with several clinical manifestations including nyctalopia, decreased visual field and decreased visual acuity. Voretigene neparvovec-rzyl uses a non-pathogenic recombinant adeno-associated virus vector serotype 2 (AAV2) to deliver cDNA encoding RPE65 protein to target cells in the retina. Voretigene neparvovec-rzyl is administered to each eye via subretinal injection. The administration of voretigene neparvovec-rzyl is recommended to be performed to each eye on separate days within a close interval. Prescribing information recommends an immunomodulatory regimen concomitant with administration, with the actual regimen dependent upon the dosing center.

This post authorization safety study will focus on further characterizing the long-term safety profile of voretigene neparvovec-rzyl in patients with RPE65 mutation-associated retinal dystrophy using an observational, longitudinal design.

ELIGIBILITY:
Inclusion Criteria:

1. Received voretigene neparvovec-rzyl in at least one eye.
2. Signed informed consent/assent (when applicable). These are obtained as required under institutional policies and applicable laws and regulations unless a consent waiver is obtained from the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).

Exclusion Criteria:

1. Previously participated in, or are currently participating in, a Spark Therapeutics clinical trial and received voretigene neparvovec-rzyl in both eyes.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who received voretigene neparvovec-rzyl in at least one eye.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Collection of all Adverse Events and Serious Adverse Events | up to 5 years
  adverse events

SECONDARY OUTCOMES:
Collection of Pregnancy Outcomes | Up to 5 years
  Follow pregnancy outcomes in participants (and female partners of male participants) who received voretigene neparvovec

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Ophthalmic Lead, Study Director — Spark Therapeutics, Inc.
Locations (10):
- United States (10):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Massachusetts Eye and Ear Institute, Boston, Massachusetts
  - Kellogg Eye Center, Ann Arbor, Michigan
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Cullen Eye Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No